CLINICAL TRIAL: NCT04214808
Title: A Randomized, Open-label, Single-dose, Crossover Study to Evaluate the Pharmacokinetics and Safety of AD-208
Brief Title: To Evaluate the Pharmacokinetics and Safety of AD-208
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-208PK
Record Dates: First submitted 2019-12-26; First posted 2020-01-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avodart Soft Capsule 0.5mg to AD-208 (Experimental): Period 1: Avodart Soft Capsule 0.5mg, 1 Capsule Period 2: AD-208, 1 tab
  Interventions: Drug: AD-208; Drug: Avodart Soft Capsule 0.5mg
- AD-208 to Avodart Soft Capsule 0.5mg (Experimental): Period 1: AD-208, 1 tab Period 2: Avodart Soft Capsule 0.5mg, 1 Capsule
  Interventions: Drug: AD-208; Drug: Avodart Soft Capsule 0.5mg

INTERVENTIONS:
Drug: AD-208 — Dutasteride 0.2mg
Drug: Avodart Soft Capsule 0.5mg — Dutasteride 0.5mg

SUMMARY:
To evaluate pharmacokinetics and safety of AD-208.

DETAILED DESCRIPTION:
The purpose is that pharmacokinetics and safety of AD-208 in healthy adult male volunteers are evaluated as compared to Avodart Soft Capsule 0.5mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Adult aged between 19 to 50 at the time of screening visit
* Weight over 50kg and Body mass index (BMI) between 17.5 kg/m2 and 30.5 kg/m2 at the time of screening visit
* No evidence of medical symptoms or signs of congenital or no chronic disease

Exclusion Criteria:

* If having a clinically significant disease or medical history for blood/tumor, genitourinary systen, liver/biliary system, kidney, respiratory system, alimentary system, endocrine system, immune system, cardiovascular system, nervous system, skin and psychical disorder, etc

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve in time plot (AUCt) | Pre-dose(0 hour) to 72 hour
  AUCt of the total ingredient of dutasteride
Peak Plasma Concentration (Cmax) | Pre-dose(0 hour) to 72 hour
  Cmax of the total ingredient of dutasteride

SECONDARY OUTCOMES:
Area under the curve in time plot (AUCinf) | Pre-dose(0 hour) to 72 hour
  AUCinf of the total ingredient of dutasteride
Time to reach Cmax(Tmax) | Pre-dose(0 hour) to 72 hour
  Tmax of the total ingredient of dutasteride
Effective half-life(t1/2) | Pre-dose(0 hour) to 72 hour
  t1/2 of the total ingredient of dutasteride
Clearance(CL/F) | Pre-dose(0 hour) to 72 hour
  CL/F of the total ingredient of dutasteride
Volume of distribution(Vd/F) | Pre-dose(0 hour) to 72 hour
  Vd/F of the total ingredient of dutasteride

OTHER OUTCOMES:
Number of participants with adverse events | From Day -1 until Day 59
  Incidence rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, M.D., Ph.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No